CLINICAL TRIAL: NCT00118898
Title: A Phase IIIB, Randomized Trial of Open-Label Efavirenz or Atazanavir With Ritonavir in Combination With Double-Blind Comparison of Emtricitabine/Tenofovir or Abacavir/Lamivudine in Antiretroviral-Naive Subjects
Brief Title: Efavirenz or Atazanavir/Ritonavir Given With Emtricitabine/Tenofovir Disoproxil Fumarate or Abacavir/Lamivudine in HIV Infected Treatment-Naive Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5202; 1U01AI068636 (NIH); ACTG 5224s (Other: Substudy)
Record Dates: First submitted 2005-07-07; First posted 2005-07-12 (Estimated); Results first posted 2011-01-10 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-09

CONDITIONS: HIV Infections
Keywords: Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — abacavir, lamivudine drug combination; Atazanavir Sulfate; efavirenz; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Ritonavir; abacavir; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- EFV, FTC/TDF, and placebo ABC/3TC (Experimental): Participants will receive EFV, FTC/TDF, and placebo for ABC/3TC for at least 96 weeks
  Interventions: Drug: Efavirenz; Drug: Emtricitabine/Tenofovir disoproxil fumarate; Drug: Abacavir/Lamivudine placebo
- EFV, ABC/3TC and placebo FTC/TDF (Experimental): Participants will receive EFV, ABC/3TC, and placebo for FTC/TDF for at least 96 weeks
  Interventions: Drug: Abacavir/Lamivudine; Drug: Efavirenz; Drug: Emtricitabine/Tenofovir disoproxil fumarate placebo
- RTV-boosted ATV, FTC/TDF, and placebo ABC/3TC (Experimental): Participants will receive RTV-boosted ATV, FTC/TDF, and placebo for ABC/3TC for at least 96 weeks
  Interventions: Drug: Atazanavir; Drug: Emtricitabine/Tenofovir disoproxil fumarate; Drug: Ritonavir; Drug: Abacavir/Lamivudine placebo
- RTV-boosted ATV, ABC/3TC, and placebo FTC/TDF (Experimental): Participants will receive RTV-boosted ATV, ABC/3TC, and placebo for FTC/TDF for at least 96 weeks
  Interventions: Drug: Abacavir/Lamivudine; Drug: Atazanavir; Drug: Ritonavir; Drug: Emtricitabine/Tenofovir disoproxil fumarate placebo

INTERVENTIONS:
Drug: Abacavir/Lamivudine — 600 mg abacavir/300 mg lamivudine tablet taken orally daily
  Other Names: ABC/3TC
  Arms: EFV, ABC/3TC and placebo FTC/TDF; RTV-boosted ATV, ABC/3TC, and placebo FTC/TDF
Drug: Atazanavir — 300 mg tablet taken orally daily
  Other Names: ATV
  Arms: RTV-boosted ATV, ABC/3TC, and placebo FTC/TDF; RTV-boosted ATV, FTC/TDF, and placebo ABC/3TC
Drug: Efavirenz — 600 mg tablet taken orally daily
  Other Names: EFV
  Arms: EFV, ABC/3TC and placebo FTC/TDF; EFV, FTC/TDF, and placebo ABC/3TC
Drug: Emtricitabine/Tenofovir disoproxil fumarate — 200 mg emtricitabine/300 mg tenofovir disoproxil fumarate tablet taken orally daily
  Other Names: FTC/TDF
  Arms: EFV, FTC/TDF, and placebo ABC/3TC; RTV-boosted ATV, FTC/TDF, and placebo ABC/3TC
Drug: Ritonavir — 100 mg tablet taken orally daily
  Other Names: RTV
  Arms: RTV-boosted ATV, ABC/3TC, and placebo FTC/TDF; RTV-boosted ATV, FTC/TDF, and placebo ABC/3TC
Drug: Abacavir/Lamivudine placebo — Placebo tablet taken orally daily
  Other Names: ABC/3TC placebo
  Arms: EFV, FTC/TDF, and placebo ABC/3TC; RTV-boosted ATV, FTC/TDF, and placebo ABC/3TC
Drug: Emtricitabine/Tenofovir disoproxil fumarate placebo — Placebo tablet taken orally daily
  Other Names: FTC/TDF placebo
  Arms: EFV, ABC/3TC and placebo FTC/TDF; RTV-boosted ATV, ABC/3TC, and placebo FTC/TDF

SUMMARY:
Currently, the preferred anti-HIV regimens used in the United States consist of two nucleoside reverse transcriptase inhibitors (NRTIs) and the nonnucleoside reverse transcriptase inhibitor (NNRTI) efavirenz (EFV). However, with new anti-HIV drugs being approved, alternative regimens need to be tested to determine if new drug combinations have increased effectiveness in treating HIV. The purpose of this study is to test the safety, tolerability, and effectiveness of four different regimens in HIV-infected adults who have never taken anti-HIV drugs.

DETAILED DESCRIPTION:
Antiretroviral (ARV) treatment regimens consisting of EFV and two NRTIs are the most commonly prescribed regimens for the initial therapy of HIV-infected people in the United States. Such regimens are popular because the drugs are easy to administer, have overall excellent efficacy, and are well tolerated. However, because of concerns about long-term drug toxicity, the development of drug resistance, and potential complications in pregnant women, it is imperative that other drug combinations be investigated as possible alternative initial regimens. Drugs recently approved by the Food and Drug Administration (FDA) for HIV treatment include the protease inhibitor (PI) atazanavir (ATV) and the two NRTI coformulations emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) and abacavir/lamivudine (ABC/3TC). Data are limited on the efficacy of these new drugs when part of anti-HIV drug regimens. This study will evaluate and compare the safety, tolerability, and efficacy of four different treatment regimens in HIV-infected treatment-naive adults.

The treatment portion of this study will last 96 weeks after the last participant is enrolled. Participants will be randomly assigned to one of four arms:

* Arm 1 participants will receive EFV, FTC/TDF, and placebo for ABC/3TC.
* Arm 2 participants will receive EFV, ABC/3TC, and placebo for FTC/TDF.
* Arm 3 participants will receive ritonavir (RTV)-boosted ATV, FTC/TDF, and placebo for ABC/3TC.
* Arm 4 participants will receive RTV-boosted ATV, ABC/3TC and placebo for FTC/TDF.

NOTE: Lopinavir/ritonavir may be used in substitution of other drugs for certain participants.

Study visits will occur at study entry; Weeks 1, 2, 4, 8, 16, and 24; and every 12 weeks thereafter. A physical exam, blood collection, and urine collection will occur at most visits. Two pharmacokinetic blood samples will be collected from participants between Weeks 4 and 24. Participants will undergo adherence training at study entry and will be asked to complete adherence questionnaires at selected study visits. Some participants will be asked to participate in ACTG A5224s, a metabolic substudy of ACTG A5202.

The Data Safety Monitoring Board (DSMB) for A5202 met in January 2008 to review the study. After reviewing the study information, the DSMB noted that certain study regimens were significantly less effective than others. Specifically, ABC/3TC-containing regimens were not as effective in controlling the virus as TDF/FTC-containing regimens for participants entering the study with high viral loads. The DSMB also commented that participants assigned to ABC/3TC had a shorter time until they experienced side effects than participants assigned to TDF/FTC. The DSMB had no safety concerns for the other drug comparisons.

Based on DSMB review, in Feb 2008 participants who started the study with high viral loads were told whether they were taking ABC/3TC or TDF/FTC and offered the option to continue or change their NRTI study drug component, after discussion with their doctor. For participants who started the study with lower screening viral loads, study treatment continued without change.

For 74 participant the reason for first treatment modification was "unblinded and switched" as a consequence of the DSMB results (33 on EFV, ABC/3TC, and placebo FTC/TDF arm; 1 on RTV-boosted ATV, FTC/TDF, and placebo ABC/3TC arm; and 40 on RTV-boosted ATV, ABC/3TC, and placebo FTC/TDF arm).

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected. A resistance assay must be obtained if the participant has evidence of recent infection. More information on this criterion can be found in the protocol.
* Antiretroviral naive, defined as 7 days or less of ARV treatment at any time prior to study entry. Participants who have received ARVs as part of postexposure prophylaxis or who have received an investigational drug that was not an NRTI, NNRTI, or PI are eligible for this study.
* HIV viral load greater than 1,000 copies/ml within 90 days prior to study entry
* Certain laboratory values obtained within 30 days prior to study entry. More information on this criterion can be found in the protocol
* Willing to use acceptable forms of contraception
* Parent or guardian able and willing to provide written informed consent, if applicable
* Hepatitis B surface antigen (HBsAg) negative at study entry

Exclusion Criteria:

* Immunomodulators (e.g., interleukins, interferons, cyclosporine), HIV vaccine, systemic cytotoxic chemotherapy, or investigational therapy within 30 days prior to study entry. Individuals receiving either stable physiologic glucocorticoid doses, corticosteroids for acute therapy for pneumocystis pneumonia, or a short course (2 weeks or less) of pharmacologic glucocorticoid therapy will not be excluded.
* Known allergy/sensitivity to study drugs or their formulations
* Active alcohol or drug use that, in the opinion of the investigator, would interfere with adherence to study requirements
* Serious illness requiring systemic treatment or hospitalization. Patients who have completed therapy or are clinically stable on therapy for at least 7 days prior to study entry are not excluded.
* Known clinically relevant cardiac conduction system disease
* Requirement for any current medications that are prohibited with any study treatment.
* Evidence of any major drug resistance-associated mutation on any genotype or evidence of significant resistance on any phenotype performed at any time prior to study entry.
* Current imprisonment or involuntary incarceration for psychiatric or physical (e.g., infectious disease) illness
* Breastfeeding. Women who become pregnant during the study will be unblinded and required to permanently discontinue their study regimens.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1864 (Actual)
Dates: Start 2005-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Daar, MD, Study Chair — Harbor-UCLA Medical Center, Los Angeles Biomedical Research Institute; Paul Sax, MD, Study Chair — Division of Infectious Diseases, Brigham and Women's Hospital
Locations (52):
- United States (51):
  - Usc Crs (1201), Los Angeles, California
  - UCLA CARE Center CRS (601), Los Angeles, California
  - Stanford CRS (501), Palo Alto, California
  - Ucsd, Avrc Crs (701), San Diego, California
  - Ucsf Aids Crs (801), San Francisco, California
  - San Mateo County AIDS Program (505), Stanford, California
  - Willow Clinic (507), Stanford, California
  - Harbor-UCLA Med. Ctr. CRS (603), Torrance, California
  - University of Colorado Hospital CRS (6101), Aurora, Colorado
  - Georgetown University CRS (GU CRS) (1008), Washington D.C., District of Columbia
  - University of Miami AIDS CRS (901), Miami, Florida
  - Emory University, Atlanta, Georgia
  - The Ponce de Leon Center CRS (5802), Atlanta, Georgia
  - Northwestern University CRS (2701), Chicago, Illinois
  - Cook County Hospital Core Center (2705), Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS (2702), Chicago, Illinois
  - Indiana University Hospital (2601), Indianapolis, Indiana
  - Wishard Hospital (2603), Indianapolis, Indiana
  - Univ of Iowa Hosp and Clinic (1504), Iowa City, Iowa
  - IHV Baltimore Treatment CRS (4651), Baltimore, Maryland
  - Johns Hopkins Adult AIDS CRS (201), Baltimore, Maryland
  - Massachusetts General Hospital ACTG CRS (101), Boston, Massachusetts
  - Brigham and Women's Hosp. ACTG CRS (107), Boston, Massachusetts
  - Bmc Actg Crs (104), Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS (103), Boston, Massachusetts
  - Washington U CRS (2101), St Louis, Missouri
  - SUNY - Buffalo (Rochester) (1102), Buffalo, New York
  - Cornell CRS (7804), New York, New York
  - Weill Med. College of Cornell Univ., The Cornell CTU -Chelsea (7803), New York, New York
  - NY Univ. HIV/AIDS CRS (401), New York, New York
  - HIV Prevention & Treatment CRS (30329), New York, New York
  - Harlem ACTG CRS (31483), New York, New York
  - AIDS Community Health Ctr. ACTG CRS (1108), Rochester, New York
  - University of Rochester ACTG CRS (1101), Rochester, New York
  - Unc Aids Crs (3201), Chapel Hill, North Carolina
  - Wake County Department of Health (30076), Chapel Hill, North Carolina
  - Duke University Medical Center Adult CRS (1601), Durham, North Carolina
  - Moses H. Cone Memorial Hospital CRS (3203), Greensboro, North Carolina
  - University of Cincinnati CRS (2401), Cincinnati, Ohio
  - Case CRS (2501), Cleveland, Ohio
  - Metro Health CRS (2503), Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS (2301), Columbus, Ohio
  - Presbyterian Medical Center - Univ. of PA (6206), Norristown, Pennsylvania
  - Hosp. of the Univ. of Pennsylvania CRS (6201), Philadelphia, Pennsylvania
  - Pitt CRS (1001), Pittsburgh, Pennsylvania
  - The Miriam Hosp. ACTG CRS (2951), Providence, Rhode Island
  - Vanderbilt Therapeutics CRS (3652), Nashville, Tennessee
  - Peabody Health Center CRS (31443), Dallas, Texas
  - University of Texas, Galveston (6301), Galveston, Texas
  - University of Washington AIDS CRS (1401), Seattle, Washington
  - University of Washington General Clinical Research (1403), Seattle, Washington
- Puerto Rico-AIDS CRS (5401), San Juan, Puerto Rico

REFERENCES:
- [Background] Anderson PL. Pharmacologic perspectives for once-daily antiretroviral therapy. Ann Pharmacother. 2004 Nov;38(11):1924-34. doi: 10.1345/aph.1E036. Epub 2004 Oct 12. PMID 15479772
- [Background] Kress KD. HIV update: emerging clinical evidence and a review of recommendations for the use of highly active antiretroviral therapy. Am J Health Syst Pharm. 2004 Oct 1;61 Suppl 3:S3-14; quiz S15-6. doi: 10.1093/ajhp/61.suppl_3.S3. PMID 15503932
- [Background] Robbins GK, De Gruttola V, Shafer RW, Smeaton LM, Snyder SW, Pettinelli C, Dube MP, Fischl MA, Pollard RB, Delapenha R, Gedeon L, van der Horst C, Murphy RL, Becker MI, D'Aquila RT, Vella S, Merigan TC, Hirsch MS; AIDS Clinical Trials Group 384 Team. Comparison of sequential three-drug regimens as initial therapy for HIV-1 infection. N Engl J Med. 2003 Dec 11;349(24):2293-303. doi: 10.1056/NEJMoa030264. PMID 14668455
- [Background] Shafer RW, Smeaton LM, Robbins GK, De Gruttola V, Snyder SW, D'Aquila RT, Johnson VA, Morse GD, Nokta MA, Martinez AI, Gripshover BM, Kaul P, Haubrich R, Swingle M, McCarty SD, Vella S, Hirsch MS, Merigan TC; AIDS Clinical Trials Group 384 Team. Comparison of four-drug regimens and pairs of sequential three-drug regimens as initial therapy for HIV-1 infection. N Engl J Med. 2003 Dec 11;349(24):2304-15. doi: 10.1056/NEJMoa030265. PMID 14668456
- [Derived] Cardone KM, Dudek S, Keat K, Bradford Y, Cindi Z, Daar ES, Gulick R, Riddler SA, Lennox JL, Sinxadi P, Haas DW, Ritchie MD. Lymphocyte Count Derived Polygenic Score and Interindividual Variability in CD4 T-cell Recovery in Response to Antiretroviral Therapy. Pac Symp Biocomput. 2024;29:594-610. PMID 38160309
- [Derived] Li B, Veturi Y, Verma A, Bradford Y, Daar ES, Gulick RM, Riddler SA, Robbins GK, Lennox JL, Haas DW, Ritchie MD. Tissue specificity-aware TWAS (TSA-TWAS) framework identifies novel associations with metabolic, immunologic, and virologic traits in HIV-positive adults. PLoS Genet. 2021 Apr 26;17(4):e1009464. doi: 10.1371/journal.pgen.1009464. eCollection 2021 Apr. PMID 33901188
- [Derived] Leonard MA, Cindi Z, Bradford Y, Bourgi K, Koethe J, Turner M, Norwood J, Woodward B, Erdem H, Basham R, Baker P, Rebeiro PF, Sterling TR, Hulgan T, Daar ES, Gulick R, Riddler SA, Sinxadi P, Ritchie MD, Haas DW. Efavirenz Pharmacogenetics and Weight Gain Following Switch to Integrase Inhibitor-Containing Regimens. Clin Infect Dis. 2021 Oct 5;73(7):e2153-e2163. doi: 10.1093/cid/ciaa1219. PMID 32829410
- [Derived] Bednasz CJ, Venuto CS, Ma Q, Daar ES, Sax PE, Fischl MA, Collier AC, Smith KY, Tierney C, Acosta EP, Mager DE, Morse GD; AIDS Clinical Trials Group Study A5202 Team. Race/Ethnicity and Protease Inhibitor Use Influence Plasma Tenofovir Exposure in Adults Living with HIV-1 in AIDS Clinical Trials Group Study A5202. Antimicrob Agents Chemother. 2019 Mar 27;63(4):e01638-18. doi: 10.1128/AAC.01638-18. Print 2019 Apr. PMID 30642925
- [Derived] Longenecker CT, Kitch D, Sax PE, Daar ES, Tierney C, Gupta SK, McComsey GA; AIDS Clinical Trials Group Study A5224s Team. Reductions in Plasma Cystatin C After Initiation of Antiretroviral Therapy Are Associated With Reductions in Inflammation: ACTG A5224s. J Acquir Immune Defic Syndr. 2015 Jun 1;69(2):168-77. doi: 10.1097/QAI.0000000000000557. PMID 26009829
- [Derived] Mollan KR, Smurzynski M, Eron JJ, Daar ES, Campbell TB, Sax PE, Gulick RM, Na L, O'Keefe L, Robertson KR, Tierney C. Association between efavirenz as initial therapy for HIV-1 infection and increased risk for suicidal ideation or attempted or completed suicide: an analysis of trial data. Ann Intern Med. 2014 Jul 1;161(1):1-10. doi: 10.7326/M14-0293. PMID 24979445
- [Derived] Sax PE, Zolopa A, Brar I, Elion R, Ortiz R, Post F, Wang H, Callebaut C, Martin H, Fordyce MW, McCallister S. Tenofovir alafenamide vs. tenofovir disoproxil fumarate in single tablet regimens for initial HIV-1 therapy: a randomized phase 2 study. J Acquir Immune Defic Syndr. 2014 Sep 1;67(1):52-8. doi: 10.1097/QAI.0000000000000225. PMID 24872136
- [Derived] Erlandson KM, Kitch D, Tierney C, Sax PE, Daar ES, Melbourne KM, Ha B, McComsey GA. Impact of randomized antiretroviral therapy initiation on glucose metabolism. AIDS. 2014 Jun 19;28(10):1451-61. doi: 10.1097/QAD.0000000000000266. PMID 24637543
- [Derived] Erlandson KM, Kitch D, Tierney C, Sax PE, Daar ES, Tebas P, Melbourne K, Ha B, Jahed NC, McComsey GA. Weight and lean body mass change with antiretroviral initiation and impact on bone mineral density. AIDS. 2013 Aug 24;27(13):2069-79. doi: 10.1097/QAD.0b013e328361d25d. PMID 24384588
- [Derived] Smith KY, Tierney C, Mollan K, Venuto CS, Budhathoki C, Ma Q, Morse GD, Sax P, Katzenstein D, Godfrey C, Fischl M, Daar ES, Collier AC; AIDS Clinical Trials Group 5202 Study Team. Outcomes by sex following treatment initiation with atazanavir plus ritonavir or efavirenz with abacavir/lamivudine or tenofovir/emtricitabine. Clin Infect Dis. 2014 Feb;58(4):555-63. doi: 10.1093/cid/cit747. Epub 2013 Nov 18. PMID 24253247
- [Derived] McComsey GA, Daar ES, O'Riordan M, Collier AC, Kosmiski L, Santana JL, Fichtenbaum CJ, Fink H, Sax PE, Libutti DE, Gerschenson M. Changes in fat mitochondrial DNA and function in subjects randomized to abacavir-lamivudine or tenofovir DF-emtricitabine with atazanavir-ritonavir or efavirenz: AIDS Clinical Trials Group study A5224s, substudy of A5202. J Infect Dis. 2013 Feb 15;207(4):604-11. doi: 10.1093/infdis/jis720. Epub 2012 Nov 29. PMID 23204164
- [Derived] Mollan K, Daar ES, Sax PE, Balamane M, Collier AC, Fischl MA, Lalama CM, Bosch RJ, Tierney C, Katzenstein D; AIDS Clinical Trials Group Study A5202 Team. HIV-1 amino acid changes among participants with virologic failure: associations with first-line efavirenz or atazanavir plus ritonavir and disease status. J Infect Dis. 2012 Dec 15;206(12):1920-30. doi: 10.1093/infdis/jis613. Epub 2012 Nov 12. PMID 23148287
- [Derived] McComsey GA, Kitch D, Sax PE, Tebas P, Tierney C, Jahed NC, Myers L, Melbourne K, Ha B, Daar ES. Peripheral and central fat changes in subjects randomized to abacavir-lamivudine or tenofovir-emtricitabine with atazanavir-ritonavir or efavirenz: ACTG Study A5224s. Clin Infect Dis. 2011 Jul 15;53(2):185-96. doi: 10.1093/cid/cir324. PMID 21690627
- [Derived] McComsey GA, Kitch D, Daar ES, Tierney C, Jahed NC, Tebas P, Myers L, Melbourne K, Ha B, Sax PE. Bone mineral density and fractures in antiretroviral-naive persons randomized to receive abacavir-lamivudine or tenofovir disoproxil fumarate-emtricitabine along with efavirenz or atazanavir-ritonavir: Aids Clinical Trials Group A5224s, a substudy of ACTG A5202. J Infect Dis. 2011 Jun 15;203(12):1791-801. doi: 10.1093/infdis/jir188. PMID 21606537
- [Derived] Daar ES, Tierney C, Fischl MA, Sax PE, Mollan K, Budhathoki C, Godfrey C, Jahed NC, Myers L, Katzenstein D, Farajallah A, Rooney JF, Pappa KA, Woodward WC, Patterson K, Bolivar H, Benson CA, Collier AC; AIDS Clinical Trials Group Study A5202 Team. Atazanavir plus ritonavir or efavirenz as part of a 3-drug regimen for initial treatment of HIV-1. Ann Intern Med. 2011 Apr 5;154(7):445-56. doi: 10.7326/0003-4819-154-7-201104050-00316. Epub 2011 Feb 14. PMID 21320923
- [Derived] Sax PE, Tierney C, Collier AC, Fischl MA, Mollan K, Peeples L, Godfrey C, Jahed NC, Myers L, Katzenstein D, Farajallah A, Rooney JF, Ha B, Woodward WC, Koletar SL, Johnson VA, Geiseler PJ, Daar ES; AIDS Clinical Trials Group Study A5202 Team. Abacavir-lamivudine versus tenofovir-emtricitabine for initial HIV-1 therapy. N Engl J Med. 2009 Dec 3;361(23):2230-40. doi: 10.1056/NEJMoa0906768. Epub 2009 Dec 1. PMID 19952143

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited at AIDS Clinical Trials Units in the United States and Puerto Rico. Recruitment occurred between September 21, 2005 (date first subject was randomized) and November 20, 2007 (date last subject was randomized).
Pre-assignment Details: 1864 were randomized. Results reported for 1857 eligible participants; 7 were subsequently found ineligible and excluded from all analyses.
Groups:
- EFV, Placebo FTC/TDF, and ABC/3TC: Participants will receive EFV, placebo for FTC/TDF, and ABC/3TC for at least 96 weeks
- RTV-boosted ATV, Placebo FTC/TDF, and ABC/3TC: Participants will receive RTV-boosted ATV, placebo for FTC/TDF, and ABC/3TC for at least 96 weeks
Period: Overall Study
Arm/Group | EFV, FTC/TDF, and Placebo ABC/3TC | EFV, Placebo FTC/TDF, and ABC/3TC | RTV-boosted ATV, FTC/TDF, and Placebo ABC/3TC | RTV-boosted ATV, Placebo FTC/TDF, and ABC/3TC
Started | 464 | 465 | 465 | 463
Initiated Treatment | 461 | 461 | 464 | 462
Completed | 343 | 324 | 342 | 322
Not Completed | 121 | 141 | 123 | 141
Not completed — Death | 6 | 11 | 6 | 8
Not completed — Lost to Follow-up | 26 | 34 | 33 | 33
Not completed — Withdrawal by Subject | 10 | 5 | 8 | 8
Not completed — Site Closure | 33 | 31 | 28 | 37
Not completed — Severe debilitation | 1 | 4 | 6 | 4
Not completed — Not compliant with requirements | 11 | 13 | 11 | 11
Not completed — Not able to get to clinic | 34 | 43 | 31 | 40

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EFV, FTC/TDF, and Placebo ABC/3TC | EFV, Placebo FTC/TDF, and ABC/3TC | RTV-boosted ATV, FTC/TDF, and Placebo ABC/3TC | RTV-boosted ATV, Placebo FTC/TDF, and ABC/3TC | Total
Number analyzed (Participants) | 464 | 465 | 465 | 463 | 1857
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 3 | 2 | 3 | 10
  Between 18 and 65 years | 461 | 454 | 461 | 458 | 1834
  >=65 years | 1 | 8 | 2 | 2 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (9.6) | 38.4 (10.5) | 38.9 (10.4) | 38.0 (9.8) | 38.4 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 98 | 78 | 75 | 322
  Male | 393 | 367 | 387 | 388 | 1535
Race/Ethnicity, Customized [Number; unit: participants] — Race/Ethnicity is collected prior to study entry, participants may opt out of reporting.
  participants
    White Non-Hispanic | 197 | 174 | 186 | 189 | 746
    Black Non-Hispanic | 151 | 164 | 147 | 153 | 615
    Hispanic (Regardless of Race) | 104 | 106 | 111 | 108 | 429
    Asian, Pacific Islander | 5 | 8 | 12 | 7 | 32
    Native American, Alaskan Native | 4 | 5 | 3 | 2 | 14
    More than One Race | 2 | 5 | 5 | 4 | 16
    Unknown | 1 | 3 | 1 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 451 | 452 | 452 | 450 | 1805
  Puerto Rico | 13 | 13 | 13 | 13 | 52
Baseline HIV-1 RNA [Mean (Standard Deviation); unit: log10 copies/mL] — Baseline RNA is calculated as the mean of the log10 pre-entry and entry values
  log10 copies/mL | 4.7 (0.7) | 4.7 (0.7) | 4.7 (0.7) | 4.7 (0.7) | 4.7 (0.7)
Screening HIV-1 RNA [Number; unit: participants]
  <100,000 copies/mL | 265 | 266 | 265 | 264 | 1060
  >=100,000 copies/mL | 199 | 199 | 200 | 199 | 797
Baseline CD4+ count [Median (Inter-Quartile Range); unit: cells/mm3] — Baseline CD4 count is the average (mean) of 2 measures taken at pre-entry and entry visits.
  cells/mm3 | 233.5 [102.5 to 333.5] | 225 [103 to 324] | 224 [87.0 to 326.5] | 236 [71.5 to 345.5] | 229.5 [89.5 to 333.8]

OUTCOME MEASURES:

1. Primary Outcome: Time From Randomization to Virologic Failure
Description: Blood samples for determining virologic failure were obtained at visit weeks 16 and 24 , and every 12 weeks thereafter. Virologic failure was defined as a confirmed plasma HIV-1 RNA level >= 1000 copies/mL at or after 16 weeks after randomization and before 24 weeks, or >=200 copies/mL at or after 24 weeks. The 5th percentile for time to virologic failure is the time (in weeks) at which 5% of the participants have experienced virologic failure.
Time Frame: Follow-up time was variable,median follow-up was 138 weeks; see 'Amount of study follow-up' outcome for details
Population: Intention to treat: All eligible participants were included in the analysis, participants were analyzed per originally assigned regimen.
Measure: Number (95% Confidence Interval); unit: Weeks
Arm/Group | EFV, FTC/TDF, and Placebo ABC/3TC | EFV, Placebo FTC/TDF, and ABC/3TC | RTV-boosted ATV, FTC/TDF, and Placebo ABC/3TC | RTV-boosted ATV, Placebo FTC/TDF, and ABC/3TC
Number analyzed (Participants) | 464 | 465 | 465 | 463
Weeks
  5th percentile time to virologic failure | 36 [24 to 60] | 24 [16 to 24] | 24 [24 to 48] | 24 [16 to 24]
  10th percentile time to virologic failure | 96 [72 to 132] | 36 [24 to 60] | 84 [48 to 156] | 36 [24 to 60]

2. Other Pre Specified Outcome: Amount of Study Follow-up
Description: Participants were to be followed for 96 weeks after the last enrollment. Accrual was expected to take 96 weeks, thus the planned follow-up time was 96 to 192 weeks, dependent on when in the study the participant enrolled. This outcome summarizes that total amount of actual follow-up in weeks from randomization to last contact.
Time Frame: Follow-up time was variable, median follow-up was 138 weeks
Population: Intention to treat: All eligible participants are included. Participants were analyzed per originally assigned regimen.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | EFV, FTC/TDF, and Placebo ABC/3TC | EFV, Placebo FTC/TDF, and ABC/3TC | RTV-boosted ATV, FTC/TDF, and Placebo ABC/3TC | RTV-boosted ATV, Placebo FTC/TDF, and ABC/3TC
Number analyzed (Participants) | 464 | 465 | 465 | 463
Weeks | 141.4 [108 to 169] | 133.3 [101.3 to 168.0] | 141.6 [105.9 to 168.1] | 137.3 [106.0 to 169.1]

3. Other Pre Specified Outcome: Number of Participants With Virologic Failure
Description: Blood samples for determining virologic failure were obtained at 16 and 24 weeks, and every 12 weeks thereafter. Virologic failure was defined as a confirmed plasma HIV-1 RNA level >= 1000 copies/mL at or after 16 weeks and before 24 weeks or >=200 copies/mL at or after 24 weeks.
Time Frame: Follow-up time was variable, median follow-up was 138 weeks; see 'Amount of study follow-up' outcome for details
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | EFV, FTC/TDF, and Placebo ABC/3TC | EFV, Placebo FTC/TDF, and ABC/3TC | RTV-boosted ATV, FTC/TDF, and Placebo ABC/3TC | RTV-boosted ATV, Placebo FTC/TDF, and ABC/3TC
Number analyzed (Participants) | 464 | 465 | 465 | 463
participants | 57 | 72 | 57 | 83

4. Secondary Outcome: Time From Treatment Dispensation to Regimen Failure (First Occurrence of Virologic Failure or Treatment Modification)
Description: Blood samples for determining virologic failure were obtained at 16 and 24 weeks, and every 12 weeks thereafter. Virologic failure was defined as a confirmed plasma HIV-1 RNA level >= 1000 copies/mL at or after 16 weeks and before 24 weeks or >=200 copies/mL at or after 24 weeks. Treatment modification was defined as the 1st modification of the regimen, including a permanent discontinuation, switch, or substitution.
Time Frame: Follow-up time was variable,median follow-up was 138 weeks; see 'Amount of study follow-up' outcome for details
Population: Participants who initiated treatment are included in this analysis. Participants were analyzed per originally assigned regimen.
Measure: Number (95% Confidence Interval); unit: Weeks
Arm/Group | EFV, FTC/TDF, and Placebo ABC/3TC | EFV, Placebo FTC/TDF, and ABC/3TC | RTV-boosted ATV, FTC/TDF, and Placebo ABC/3TC | RTV-boosted ATV, Placebo FTC/TDF, and ABC/3TC
Number analyzed (Participants) | 461 | 461 | 464 | 462
Weeks
  5th percentile time to regimen failure | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 16] | 4 [4 to 4]
  10th percentile time to regimen failure | 16 [4 to 16] | 4 [4 to 4] | 16 [16 to 24] | 4 [4 to 16]
  25th percentile time to regimen failure | 72 [48 to 96] | 24 [16 to 36] | 84 [60 to 108] | 36 [24 to 36]

5. Secondary Outcome: The Number of Participants With HIV-1 RNA Levels Less Than 50 Copies/mL
Time Frame: At Weeks 48 and 96
Population: Intention to treat: All participants with RNA data were included, complete-case approach.
Measure: Number; unit: Participants
Arm/Group | EFV, FTC/TDF, and Placebo ABC/3TC | EFV, Placebo FTC/TDF, and ABC/3TC | RTV-boosted ATV, FTC/TDF, and Placebo ABC/3TC | RTV-boosted ATV, Placebo FTC/TDF, and ABC/3TC
Number analyzed (Participants) | 464 | 465 | 465 | 463
Participants
  Number of Participants with RNA data at Week 48 | 415 | 400 | 416 | 411
  Number with HIV-1 RNA <50 copies/ml at Week 48 | 372 | 346 | 348 | 322
  Number of Participants with RNA data at Week 96 | 379 | 361 | 384 | 374
  Number with HIV-1 RNA <50 copies/ml at Week 96 | 345 | 328 | 345 | 317

6. Secondary Outcome: Number of Participants With HIV-1 RNA Levels Less Than 200 Copies/mL
Time Frame: At Weeks 48 and 96
Population: Intention to treat: All participants with RNA data were included, complete-case approach.
Measure: Number; unit: Participants
Arm/Group | EFV, FTC/TDF, and Placebo ABC/3TC | EFV, Placebo FTC/TDF, and ABC/3TC | RTV-boosted ATV, FTC/TDF, and Placebo ABC/3TC | RTV-boosted ATV, Placebo FTC/TDF, and ABC/3TC
Number analyzed (Participants) | 464 | 465 | 465 | 463
Participants
  Number of Participants with RNA data at Week 48 | 415 | 400 | 416 | 411
  Number with HIV-1 RNA <200 copies/ml at Week 48 | 398 | 377 | 391 | 372
  Number of Participants with RNA data at Week 96 | 379 | 361 | 384 | 374
  Number with HIV-1 RNA <200 copies/ml at Week 96 | 362 | 342 | 368 | 346

7. Secondary Outcome: Change in CD4 Count (Cells/mm3) From Baseline
Description: Change was calculated as the CD4 count at Week 48 (or at Week 96) minus the baseline CD4 count (mean of pre-entry and entry values).
Time Frame: At Weeks 48 and 96
Population: Intention to treat: All participants with CD4 data were included, complete-case approach.
Measure: Median (Inter-Quartile Range); unit: Cells/mm3
Arm/Group | EFV, FTC/TDF, and Placebo ABC/3TC | EFV, Placebo FTC/TDF, and ABC/3TC | RTV-boosted ATV, FTC/TDF, and Placebo ABC/3TC | RTV-boosted ATV, Placebo FTC/TDF, and ABC/3TC
Number analyzed (Participants) | 464 | 465 | 465 | 463
Cells/mm3
  Week 48 | 163 [96.5 to 250.0] | 188 [102.5 to 277.5] | 175 [108 to 290] | 177.5 [106.0 to 275.5]
  Week 96 | 220.5 [134.5 to 323.5] | 250.5 [158.0 to 364.3] | 251.5 [165.5 to 362.5] | 250.3 [153.0 to 350.0]

8. Secondary Outcome: Number of Participants With Virologic Failure and Emergence of Major Resistance
Description: Emergence of resistant virus was assessed by genotypic testing performed at Stanford University for all participants who met criteria for virologic failure and retrospectively on baseline samples from these participants. Major mutations were defined by International AIDS Society-United States of America (2008), as well as T69D, L74I, G190C/E/Q/T/V for reverse transcriptase and L24I, F53L, I54V/A/T/S, G73C/S/T/A, N88D for protease.
Time Frame: Follow-up time was variable,median follow-up was 138 weeks; see 'Amount of study follow-up' outcome for details
Population: Intention to treat: All eligible participants are included. Participants were analyzed per originally assigned regimen.
Measure: Number; unit: participants
Arm/Group | EFV, FTC/TDF, and Placebo ABC/3TC | EFV, Placebo FTC/TDF, and ABC/3TC | RTV-boosted ATV, FTC/TDF, and Placebo ABC/3TC | RTV-boosted ATV, Placebo FTC/TDF, and ABC/3TC
Number analyzed (Participants) | 464 | 465 | 465 | 463
participants | 27 | 41 | 5 | 12

9. Secondary Outcome: Number of Participants Experiencing Certain Targeted Clinical Events, Including Death, AIDS-defining Illness, and HIV-1 Related Events.
Description: AIDS-defining illnesses were defined per CDC category C definition. HIV-1 related events were defined per CDC category B definition. Events underwent study chair review for classification. See link below for more details.
  http://www.cdc.gov/mmwr/preview/mmwrhtml/00018871.htm
Time Frame: Follow-up time was variable, median follow-up was 138 weeks; see 'Amount of study follow-up' outcome for details
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | EFV, FTC/TDF, and Placebo ABC/3TC | EFV, Placebo FTC/TDF, and ABC/3TC | RTV-boosted ATV, FTC/TDF, and Placebo ABC/3TC | RTV-boosted ATV, Placebo FTC/TDF, and ABC/3TC
Number analyzed (Participants) | 464 | 465 | 465 | 463
Participants
  Death | 6 | 11 | 6 | 8
  AIDS-defining illness | 14 | 25 | 20 | 23
  HIV-1 relatated event | 56 | 61 | 57 | 63

10. Secondary Outcome: Change in Fasting Total Cholesterol Level From Baseline
Description: Only fasting results are included. The protocol did not require that samples be collected fasting.
Time Frame: At Weeks 48 and 96
Population: Intention to treat: All participants with fasting lipids data were included, complete-case approach.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | EFV, FTC/TDF, and Placebo ABC/3TC | EFV, Placebo FTC/TDF, and ABC/3TC | RTV-boosted ATV, FTC/TDF, and Placebo ABC/3TC | RTV-boosted ATV, Placebo FTC/TDF, and ABC/3TC
Number analyzed (Participants) | 464 | 465 | 465 | 463
mg/dL
  Week 48 | 22 [2 to 43] | 35 [15.5 to 58] | 11 [-9 to 36] | 30 [9 to 54]
  Week 96 | 23 [2 to 41] | 33 [10 to 60] | 14 [-6 to 39] | 25 [7 to 50]

11. Secondary Outcome: Change in Fasting High-density Lipoprotein (HDL) Cholesterol Level From Baseline
Description: Only fasting results are included. The protocol did not require that samples be collected fasting.
Time Frame: At Weeks 48 and 96
Population: Intention to treat: All participants with fasting lipids data were included, complete-case approach.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | EFV, FTC/TDF, and Placebo ABC/3TC | EFV, Placebo FTC/TDF, and ABC/3TC | RTV-boosted ATV, FTC/TDF, and Placebo ABC/3TC | RTV-boosted ATV, Placebo FTC/TDF, and ABC/3TC
Number analyzed (Participants) | 464 | 465 | 465 | 463
mg/dL
  Week 48 | 8 [3 to 15] | 10 [4 to 18] | 5 [-2 to 10] | 8 [1 to 16]
  Week 96 | 9 [2 to 16] | 11 [3.5 to 18.5] | 4 [-1 to 11] | 7 [1 to 15]

12. Secondary Outcome: Change in Fasting Non-high Density Lipoprotein (Non-HDL) Cholesterol Level From Baseline
Description: Only fasting results are included. The protocol did not require that samples be collected fasting.
Time Frame: At Weeks 48 and 96
Population: Intention to treat: All participants with fasting lipids data were included, complete-case approach.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | EFV, FTC/TDF, and Placebo ABC/3TC | EFV, Placebo FTC/TDF, and ABC/3TC | RTV-boosted ATV, FTC/TDF, and Placebo ABC/3TC | RTV-boosted ATV, Placebo FTC/TDF, and ABC/3TC
Number analyzed (Participants) | 464 | 465 | 465 | 463
mg/dL
  Week 48 | 14 [-4.5 to 30.5] | 23 [3 to 47] | 8 [-11 to 30] | 20 [-1 to 42]
  Week 96 | 13.5 [-5.5 to 31.0] | 18 [0 to 45] | 10 [-9.5 to 34.0] | 18 [2 to 43]

13. Primary Outcome: Time From Treatment Dispensation to a Grade 3/4 Safety Event
Description: Grade 3/4 safety event is defined as a grade 3 or 4 sign, symptom, or laboratory abnormality that is at least one grade higher than at baseline, total bilirubin and creatine kinase (CPK) were excluded. Grading used the Division of AIDS (DAIDS) 2004 Severity of Adverse Events Tables.
Time Frame: All follow-up while on initially assigned regimen; the median (25th, 75th percentile) follow-up while on initial regimen was 120 (54, 156) weeks and the range was 0 to 205 weeks.
Population: As-treated: Participants who initiated treatment are included in this analysis. Follow-up while on initially assigned treatment is included in the at-risk period.
Measure: Number (95% Confidence Interval); unit: Weeks
Arm/Group | EFV, FTC/TDF, and Placebo ABC/3TC | EFV, Placebo FTC/TDF, and ABC/3TC | RTV-boosted ATV, FTC/TDF, and Placebo ABC/3TC | RTV-boosted ATV, Placebo FTC/TDF, and ABC/3TC
Number analyzed (Participants) | 461 | 461 | 464 | 462
Weeks
  5th percentile time to a grade 3/4 safety event | 2.6 [1.6 to 4.3] | 1.3 [1.0 to 1.3] | 3.0 [1.3 to 4.9] | 1.3 [1.0 to 1.7]
  10th percentile time to a grade 3/4 safety event | 7.9 [4.3 to 13.0] | 2.0 [1.3 to 3.9] | 8.1 [5.1 to 17.9] | 3.9 [1.9 to 7.1]
  25th percentile time to a grade 3/4 safety event | 59.3 [41.7 to 91.7] | 16.0 [8.3 to 22.0] | 81.4 [47.9 to 111.3] | 44.4 [24.3 to 52.1]

14. Other Pre Specified Outcome: Cumulative Probability of Not Experiencing Virologic Failure
Description: Kaplan-Meier estimate of the cumulative survival probability at week 48 and 96. Blood samples for determining virologic failure were obtained at 16 and 24 weeks, and every 12 weeks thereafter. Virologic failure was defined as a confirmed plasma HIV-1 RNA level >= 1000 copies/mL at or after 16 weeks and before 24 weeks or >=200 copies/mL at or after 24 weeks.
Time Frame: At week 48 and 96
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | EFV, FTC/TDF, and Placebo ABC/3TC | EFV, Placebo FTC/TDF, and ABC/3TC | RTV-boosted ATV, FTC/TDF, and Placebo ABC/3TC | RTV-boosted ATV, Placebo FTC/TDF, and ABC/3TC
Number analyzed (Participants) | 464 | 465 | 465 | 463
percentage of participants
  Week 48 | 94 [91 to 96] | 88 [85 to 91] | 92 [89 to 94] | 88 [84 to 90]
  Week 96 | 90 [87 to 92] | 85 [82 to 88] | 89 [86 to 92] | 83 [79 to 87]

15. Primary Outcome: Time From Treatment Dispensation to Treatment Modification
Description: Treatment modification is defined as the 1st modification of the regimen, including a permanent discontinuation, switch, or substitution.
Time Frame: Follow-up time was variable,median follow-up was 138 weeks; see 'Amount of study follow-up' outcome for details
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Weeks
Arm/Group | EFV, FTC/TDF, and Placebo ABC/3TC | EFV, Placebo FTC/TDF, and ABC/3TC | RTV-boosted ATV, FTC/TDF, and Placebo ABC/3TC | RTV-boosted ATV, Placebo FTC/TDF, and ABC/3TC
Number analyzed (Participants) | 461 | 461 | 464 | 462
Weeks
  5th percentile time to treatment modification | 3.4 [1.6 to 7.1] | 1.4 [1.3 to 1.6] | 7.9 [2.1 to 14.0] | 1.6 [1.3 to 2.4]
  10th percentile time to treatment modification | 15.0 [7.6 to 23.7] | 2.1 [1.6 to 4.1] | 24.9 [14.4 to 38.1] | 5.0 [2.6 to 12.6]
  25th percentile time to treatment modification | 83.7 [63.0 to 119.6] | 27.4 [21.7 to 34.9] | 108.9 [85.1 to 144.1] | 43.6 [30.3 to 56.0]

16. Other Pre Specified Outcome: Number of Participants With a Grade 3/4 Safety Event
Description: Grade 3/4 safety event is defined as a grade 3 or 4 sign, symptom, or laboratory abnormality that is at least one grade higher than at baseline, total bilirubin and creatine kinase (CPK) were excluded. Grading used the Division of AIDS (DAIDS) 2004 Severity of Adverse Events Tables. As-treated analysis censored at 1st modification of initially assigned regimen, participants who never started treatment were excluded.
Time Frame: Over all study follow-up while on initially assigned treatment, median follow-up was 120 weeks
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | EFV, FTC/TDF, and Placebo ABC/3TC | EFV, Placebo FTC/TDF, and ABC/3TC | RTV-boosted ATV, FTC/TDF, and Placebo ABC/3TC | RTV-boosted ATV, Placebo FTC/TDF, and ABC/3TC
Number analyzed (Participants) | 461 | 461 | 464 | 462
participants | 145 | 182 | 137 | 156

17. Other Pre Specified Outcome: Cumulative Probability of Not Experiencing a Grade 3/4 Safety Event
Description: Kaplan-Meier estimate of the cumulative survival probability at week 48 and 96. Grade 3/4 safety event is defined as a grade 3 or 4 sign, symptom, or laboratory abnormality that is at least one grade higher than at baseline, total bilirubin and creatine kinase (CPK) were excluded. Grading used the Division of AIDS (DAIDS) 2004 Severity of Adverse Events Tables. As-treated analysis censored at 1st modification of initially assigned regimen, participants who never started treatment were excluded.
Time Frame: At week 48 and 96
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | EFV, FTC/TDF, and Placebo ABC/3TC | EFV, Placebo FTC/TDF, and ABC/3TC | RTV-boosted ATV, FTC/TDF, and Placebo ABC/3TC | RTV-boosted ATV, Placebo FTC/TDF, and ABC/3TC
Number analyzed (Participants) | 461 | 461 | 464 | 462
percentage of participants
  Week 48 | 78 [73 to 81] | 64 [60 to 69] | 79 [75 to 82] | 73 [68 to 77]
  Week 96 | 70 [65 to 74] | 58 [53 to 63] | 73 [68 to 77] | 66 [61 to 70]

18. Other Pre Specified Outcome: Number of Participants With Treatment Modification
Description: as for outcome 15
Time Frame: Follow-up time was variable, median follow-up was 138 weeks; see 'Amount of study follow-up' outcome for details
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | EFV, FTC/TDF, and Placebo ABC/3TC | EFV, Placebo FTC/TDF, and ABC/3TC | RTV-boosted ATV, FTC/TDF, and Placebo ABC/3TC | RTV-boosted ATV, Placebo FTC/TDF, and ABC/3TC
Number analyzed (Participants) | 461 | 461 | 464 | 462
participants | 152 | 239 | 138 | 216

19. Other Pre Specified Outcome: Cumulative Probability of Not Experiencing Treatment Modification
Description: Kaplan-Meier estimate of the cumulative survival probability at week 48 and 96. Treatment modification is defined as the 1st modification of the regimen, including a permanent discontinuation, switch, or substitution.
Time Frame: At week 48 and 96
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | EFV, FTC/TDF, and Placebo ABC/3TC | EFV, Placebo FTC/TDF, and ABC/3TC | RTV-boosted ATV, FTC/TDF, and Placebo ABC/3TC | RTV-boosted ATV, Placebo FTC/TDF, and ABC/3TC
Number analyzed (Participants) | 461 | 461 | 464 | 462
percentage of participants
  Week 48 | 80 [76 to 84] | 67 [63 to 71] | 86 [82 to 89] | 73 [69 to 77]
  Week 96 | 73 [69 to 77] | 56 [52 to 61] | 77 [73 to 81] | 62 [58 to 66]

20. Other Pre Specified Outcome: Number of Participants With Regimen Failure
Description: as for outcome 4
Time Frame: Follow-up time was variable, median follow-up was 138 weeks; see 'Amount of study follow-up' outcome for details
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | EFV, FTC/TDF, and Placebo ABC/3TC | EFV, Placebo FTC/TDF, and ABC/3TC | RTV-boosted ATV, FTC/TDF, and Placebo ABC/3TC | RTV-boosted ATV, Placebo FTC/TDF, and ABC/3TC
Number analyzed (Participants) | 461 | 461 | 464 | 462
participants | 162 | 246 | 157 | 233

21. Other Pre Specified Outcome: Cumulative Probability of Not Experiencing Regimen Failure
Description: Kaplan-Meier estimate of the cumulative survival probability at week 48 and 96. Blood samples for determining virologic failure were obtained at 16 and 24 weeks, and every 12 weeks thereafter. Virologic failure was defined as a confirmed plasma HIV-1 RNA level >= 1000 copies/mL at or after 16 weeks and before 24 weeks or >=200 copies/mL at or after 24 weeks. Treatment modification was defined as the 1st modification of the regimen, including a permanent discontinuation, switch, or substitution.
Time Frame: At week 48 and 96
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | EFV, FTC/TDF, and Placebo ABC/3TC | EFV, Placebo FTC/TDF, and ABC/3TC | RTV-boosted ATV, FTC/TDF, and Placebo ABC/3TC | RTV-boosted ATV, Placebo FTC/TDF, and ABC/3TC
Number analyzed (Participants) | 461 | 461 | 464 | 462
percentage of participants
  Week 48 | 79 [75 to 82] | 64 [59 to 68] | 80 [76 to 84] | 66 [62 to 70]
  Week 96 | 70 [66 to 74] | 54 [49 to 58] | 73 [69 to 77] | 57 [52 to 61]

22. Secondary Outcome: Change in Fasting Triglyceride Level From Baseline
Description: Only fasting results are included. The protocol did not require that samples be collected fasting.
Time Frame: At Weeks 48 and 96
Population: Intention to treat: All participants with fasting lipids data were included, complete-case approach.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | EFV, FTC/TDF, and Placebo ABC/3TC | EFV, Placebo FTC/TDF, and ABC/3TC | RTV-boosted ATV, FTC/TDF, and Placebo ABC/3TC | RTV-boosted ATV, Placebo FTC/TDF, and ABC/3TC
Number analyzed (Participants) | 464 | 465 | 465 | 463
mg/dL
  Week 48 | 10 [-29 to 44] | 15 [-20 to 65] | 14 [-18 to 52] | 24 [-12 to 80]
  Week 96 | 9 [-27 to 48] | 14 [-22 to 54] | 11 [-21 to 47] | 33 [-9 to 78]

ADVERSE EVENTS:
Time Frame: From treatment dispensation until off-study, participant follow-up time was variable. Median follow-up was 138 weeks, see 'Amount of study follow-up' for more details.
Description: Grade≥2 CNS, nausea, diarrhea & other Grade>3 signs/symptoms (S/Sx). Diagnoses per ACTG criteria for clinical events & diseases. All Creatinine, bilirubin, fasting lipid & glucose, and other Grade>3 labs. All S/Sx or labs that lead to a change in study treatment. See DAIDS Grading Severity of AEs, V1.0, Dec04, http://rcc.tech-res-intl.com
Arm/Group | EFV, FTC/TDF, and Placebo ABC/3TC | EFV, Placebo FTC/TDF, and ABC/3TC | RTV-boosted ATV, FTC/TDF, and Placebo ABC/3TC | RTV-boosted ATV, Placebo FTC/TDF, and ABC/3TC
Serious Adverse Events (participants affected / at risk) | 48/461 | 62/461 | 58/464 | 71/462
Other Adverse Events (participants affected / at risk) | 434/461 | 433/461 | 453/464 | 461/462
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EFV, FTC/TDF, and Placebo ABC/3TC (N=461) | EFV, Placebo FTC/TDF, and ABC/3TC (N=461) | RTV-boosted ATV, FTC/TDF, and Placebo ABC/3TC (N=464) | RTV-boosted ATV, Placebo FTC/TDF, and ABC/3TC (N=462)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 3 | 0 | 1
Accidental death (General disorders) | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 0 | 0 | 0
Adenomyosis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Adverse drug reaction (General disorders) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2 | 0 | 2
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 0
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 14 | 5
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Blood triglycerides (Investigations) | 0 | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 2 | 4 | 0 | 2
Burkitt's lymphoma (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Cardio-respiratory arrest (General disorders) | 0 | 0 | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 3 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 2 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 0
Death (General disorders) | 1 | 5 | 1 | 2
Demyelinating polyneuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression suicidal (Psychiatric disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 5 | 2 | 7
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
HIV infection (Infections and infestations) | 0 | 0 | 2 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 2
Hepatitis C (Infections and infestations) | 0 | 1 | 0 | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 13 | 14
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 3 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Inflammatory carcinoma of the breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 1 | 3 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 3 | 1 | 0
Liver function test abnormal (Investigations) | 1 | 1 | 1 | 3
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Lung infection pseudomonal (Infections and infestations) | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0
Meningitis cryptococcal (Infections and infestations) | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Multiple drug overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Mycobacterium avium complex infection (Infections and infestations) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Narcotic intoxication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 3 | 1
Neurotoxicity (Nervous system disorders) | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Ovarian mass (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Personality change (Psychiatric disorders) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 3 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Status epilepticus (Nervous system disorders) | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 2 | 3 | 0 | 1
Suicide attempt (Psychiatric disorders) | 3 | 2 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Transaminases increased (Investigations) | 2 | 0 | 0 | 0
Transient global amnesia (Nervous system disorders) | 0 | 0 | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 1 | 0 | 0 | 0
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EFV, FTC/TDF, and Placebo ABC/3TC (N=461) | EFV, Placebo FTC/TDF, and ABC/3TC (N=461) | RTV-boosted ATV, FTC/TDF, and Placebo ABC/3TC (N=464) | RTV-boosted ATV, Placebo FTC/TDF, and ABC/3TC (N=462)
Abnormal dreams (Psychiatric disorders) | 20 | 26 | 2 | 3
Alanine aminotransferase increased (Investigations) | 67 | 70 | 53 | 52
Aspartate aminotransferase increased (Investigations) | 73 | 67 | 63 | 61
Blood bilirubin increased (Investigations) | 47 | 57 | 412 | 430
Blood cholesterol (Investigations) | 51 | 70 | 40 | 59
Blood cholesterol abnormal (Investigations) | 220 | 282 | 179 | 267
Blood creatinine increased (Investigations) | 21 | 27 | 42 | 32
Blood glucose abnormal (Investigations) | 184 | 195 | 180 | 202
Blood glucose decreased (Investigations) | 34 | 24 | 26 | 28
Blood phosphorus decreased (Investigations) | 36 | 32 | 29 | 29
Blood sodium decreased (Investigations) | 38 | 45 | 48 | 35
Blood triglycerides (Investigations) | 25 | 49 | 18 | 46
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 23 | 15 | 27
Depression (Psychiatric disorders) | 41 | 40 | 34 | 42
Diarrhoea (Gastrointestinal disorders) | 54 | 78 | 61 | 81
Dizziness (Nervous system disorders) | 42 | 53 | 16 | 9
Drug hypersensitivity (Immune system disorders) | 22 | 49 | 29 | 30
Fatigue (General disorders) | 41 | 49 | 24 | 35
Haemoglobin decreased (Investigations) | 19 | 27 | 18 | 24
Headache (Nervous system disorders) | 37 | 41 | 29 | 42
Hypertension (Vascular disorders) | 29 | 27 | 14 | 27
Insomnia (Psychiatric disorders) | 28 | 33 | 8 | 20
Low density lipoprotein (Investigations) | 40 | 55 | 27 | 42
Low density lipoprotein abnormal (Investigations) | 188 | 228 | 156 | 205
Nausea (Gastrointestinal disorders) | 58 | 77 | 51 | 86
Neutrophil count decreased (Investigations) | 79 | 88 | 69 | 71
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 25 | 9 | 25
Platelet count decreased (Investigations) | 28 | 27 | 25 | 25
Pyrexia (General disorders) | 20 | 52 | 36 | 50
Rash (Skin and subcutaneous tissue disorders) | 17 | 26 | 18 | 25
Rash generalised (Skin and subcutaneous tissue disorders) | 10 | 29 | 9 | 20
Vomiting (Gastrointestinal disorders) | 24 | 43 | 24 | 38
White blood cell count decreased (Investigations) | 43 | 47 | 37 | 36

LIMITATIONS AND CAVEATS:
HIV-1 drug resistance testing and HLA-B*5701 testing were not standard of care during enrollment. EFV and RTV-boosted ATV were open-label, and blinded FTC/TDF vs. ABC/3TC were unblinded in the >=100,000 cp/mL screening viral load stratum Feb 2008.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less